CLINICAL TRIAL: NCT05628038
Title: Hypofractionated Radiotherapy Combined With Toripalimab and Chemotherapy +/- Target Therapy for Locally Recurrent Rectal Cancer: a Single-arm, Two-cohort, Phase II Trial (TORCH-R)
Brief Title: The Combination of Hypofractionated Radiotherapy and Immunotherapy in Locally Recurrent Rectal Cancer
Acronym: TORCH-R
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2022-289-3006
Record Dates: First submitted 2022-11-17; First posted 2022-11-28 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Recurrent Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — spartalizumab; toripalimab; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin; Irinotecan; raltitrexed; Cetuximab; Bevacizumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): The enrolled patients will receive 25-40Gy/5Fx irradiation or 15-30Gy/5Fx reirradiation (pelvic radiation history) for pelvic recurrence.
  Cohort A patients will receive CAPOX, FOLFIRI or mFOLFOX6 chemotherapy andcohort B patients will receive CAPOX, FOLFIRI, mFOLFOX6, mXELIRI, irinotecan and raltitrexed, or oxaliplatin and raltitrexed chemotherapy, based on previous chemotherapy and adverse reactions to chemotherapy agents or at the discretion of the oncologist.
  All metastasis sites will receive stereotactic ablative radiotherapy (SABR) between chemoimmunotherapy cycles. Five-fraction regimens (25-50Gy/5Fx) are delivered daily. Dose Constraints are based on SABR-COMET 10 trial.
  Besides, according to the medical oncologist recommendation, patients with unresectable pelvic recurrence or distant metastasis will receive target therapy based on the KRAS/NRAS/BRAF mutation station.
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine; Drug: 5FU; Drug: folinic acid; Drug: Oxaliplatin; Drug: Irinotecan; Drug: Raltitrexed; Drug: Cetuximab; Drug: Bevacizumab; Radiation: Radiation

INTERVENTIONS:
Drug: PD-1 antibody — PD-1 antibody (Toripalimab): 240mg q3w or 160mg q2w
  Other Names: Toripalimab
Drug: Capecitabine — Capecitabine: 1000mg/m2 d1-14 q3w
  Other Names: Xeloda
Drug: 5FU — 400 mg/m2 (bolus) and 2400 mg/m2 (continuous infusion for 48hr)
Drug: folinic acid — 400 mg/m2 q2w
Drug: Oxaliplatin — 130 mg/m² q3w or 85 mg/m² q2w
Drug: Irinotecan — 180 mg/m² q2w and 200 mg/m² q3w
Drug: Raltitrexed — 2 mg/m² q2w and 3 mg/m² q3w
Drug: Cetuximab — 400 mg/m² q2w
Drug: Bevacizumab — 5 mg/kg q2w or 7.5mg/kg q3w
Radiation: Radiation — 25-40Gy/5Fx irradiation or 15-30Gy/5Fx reirradiation (pelvic radiation history) for pelvic recurrence tumor.
  35-60Gy/5-8Fx irradiation for distance metastasis tumor.

SUMMARY:
The study is a prospective, single-center, single-arm, two-cohort, phase II clinical trial. Patients aged 18 years or older who had pelvic recurrence rectal cancer with or without resectable distant metastasis, with treatment naive disease (cohort A) or progressive disease after first-line chemotherapy (cohort B), Eastern Cooperative Oncology Group performance status of 0-1, will receive 25-40Gy/5Fx irradiation or 15-30Gy/5Fx reirradiation (pelvic radiation history), 18 weeks toripalimab and investigator's choice of chemotherapy +/- target therapy, and stereotactic ablative radiotherapy (SABR) for all metastatic lesions between chemoimmunotherapy cycles, followed by multidisciplinary team (MDT) for decision:follow-up of complete response (CR), radical surgery, sustained treatment of non resection, or exit.

The primary endpoint was local objective response rate. Secondary endpoints were extrapelvic objective response rate, R0 resection rate, duration of response, progression-free survival, overall survival, and safety and tolerability of the treatment.

Shanghai Junshi Biomedical Technology Co., Ltd. Provides the first three cycles of toripalimab for free and has purchased liability insurance for clinical trial subjects.

DETAILED DESCRIPTION:
For patients with locally recurrent rectal cancer (LRRC), response rate of chemoradiotherapy is 40-50% and only approximately 40-50% of patients with recurrent rectal cancer can undergo R0 resection. Recent studies have shown promising synergistic effects of the combination of immunotherapy (PD-1/PD-L1 antibodies) and neoadjuvant chemoradiotherapy (nCRT) in locally advanced rectal cancer (LARC). Thus, for LRRC patients, addition of immunotherapy to CRT is likely to further improve the response rate and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18-75 years old at the time of signing the informed consent form.
* ECOG performance status 0-1.
* MRI/enhanced CT confirmed pelvic recurrence. According to RECIST 1.1, there is at least one measurable pelvic lesion.
* Distant metastasis lesions are no more than 5 and metastatic organ are no more than 3.
* No prior radiotherapy within 6 month.
* Previous system therapy. Patients Group Cohort A: participants with pelvic recurrence who have not previously been treated with first-line chemotherapy. Cohort B: Patients with disease progression or new lesions after first-line chemotherapy.
* Has an investigator determined life expectancy of at least 24 weeks.
* Demonstrate adequate organ function (bone marrow, liver, kidney and clotting function) within 7 days before the first administration without using blood products or hematopoietic stimulating factors.
* Non pregnant or lactating patients. Effective contraceptive methods should be used during the study and within 6 months of the last administration.
* Fully informed and willing to provide written informed consent for the trial.

Exclusion Criteria:

* Neutrophil < 1.5×10^9/L, PLT < 100×10^9/L (PLT < 80×10^9/L in patients with liver metastasis), or Hb < 90g/L; blood transfusion within 2 weeks before enrollment is not allowed to meet the enrollment criteria.
* TBIL > 1.5 ULN, or TBIL > 2.5 ULN in patients with liver metastasis.
* AST or ALT > 2.5 ULN, or ALT and / or AST > 5 ULN in patients with liver metastasis.
* Cr > 1.5 ULN, or creatinine clearance < 50ml / min (calculated according to Cockcroft Gault formula).
* APTT > 1.5 ULN, PT > 1.5 ULN (subject to the normal value of the clinical trial research center).
* Serious electrolyte abnormalities.
* Urinary protein ≥ 2+, or 24-hour urine protein ≥1.0g/24h.
* Uncontrolled hypertension: SBP >140mmHg or DBP > 90mmHg.
* The presence of gastrointestinal diseases such as gastric or duodenal active ulcers, ulcerative colitis or unresected tumours with active bleeding; or other conditions likely to cause gastrointestinal bleeding or perforation; or unhealed gastrointestinal perforation or gastrointestinal fistula after surgical treatment.
* A history of arterial thrombosis or deep vein thrombosis within 6 months; a history of bleeding or evidence of bleeding tendency within 2 months.
* A history of heart disease within 6 months (including congestive heart failure, acute myocardial infarction, severe/unstable angina, coronary artery bypass grafting, cardiac insufficiency ≥ NYHA grade 2 and LVEF<50%).
* Uncontrolled malignant pleural effusion, ascites, or pericardial effusion.
* History of anti-PD-1, PD-L1, PD-L2, CTLA-4 or any other specific T cell co-stimulation or checkpoint pathway targeted therapy.
* The presence of a clinically detectable second primary malignancy, or history of other malignancies within 5 years excluding adequately treated non-melanoma skin cancer, carcinoma in situ of cervix and superficial bladder tumour (non-invasive tumour, or carcinoma in situ, or T1).
* A history of liver disease including, but not limited to HBV infection or HBV DNA positive(≥1×10^4/ml), HCV infection or HCV DNA positive(≥1×10^3/ml) and liver cirrhosis.
* Pregnant or lactating women or women who may be pregnant have a positive pregnancy test before the first medication; Or the female participants themselves and their partners who were unwilling to implement strict contraception during the study period.
* The investigator considers that the subject is not suitable to participate in this clinical study due to any clinical or laboratory abnormalities or compliance problems.
* Serious mental abnormalities.
* The diameter of brain metastasis is greater than 3cm or the total volume is greater than 30cc.
* Clinical or radiological evidence of spinal cord compression, or tumours within 3 mm of the spinal cord on MRI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Local objective response rate | up to 1 year
  the proportion of patients with the best pelvic response of confirmed complete or partial response according to RECIST 1.1, as assessed by the investigator.

SECONDARY OUTCOMES:
Extrapelvic objective response rate | up to 1 year
  proportion of patients with confirmed extrapelvic complete or partial response per RECIST 1.1.
R0 resection rate | up to 1 year
  the proportion of patients who achieve R0 resection of pelvic recurrent tumour after therapy.
Duration of response (DOR) | up to 1 year
  time from the first documented pelvic objective response to pelvic or extrapelvic disease progression in patients with confirmed response.
Progression-Free Survival | up to 3 year
  time from the date of start treatment until disease progression or censored at last follow-up or death.
Overall Survival | up to 3 year
  from the date of start treatment until the date of death from any cause or censored at last follow-up.
Safety and tolerability of the treatment | up to 1 year
  proportion of patients with treatment-related acute toxicities as assessed by NCI CTCAE v5.0, from treatment initiation until 90 days upon completion of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wan J, Wu R, Fu M, Shen L, Zhang H, Wang Y, Wang Y, Zhou S, Chen Y, Xia F, Zhang Z. TORCH-R trial protocol: hypofractionated radiotherapy combined with chemotherapy and toripalimab for locally recurrent rectal cancer: a prospective, single-arm, two-cohort, phase II trial. Front Oncol. 2023 Nov 20;13:1304767. doi: 10.3389/fonc.2023.1304767. eCollection 2023. PMID 38053659